CLINICAL TRIAL: NCT07301385
Title: Evaluation of Head-Mounted Spatial Computing and Three-Dimensional (3D) Visualization in Ocular Microsurgery: A Feasibility and Safety Study
Brief Title: Evaluation of Head-Mounted Spatial Computing and Three-Dimensional (3D) Visualization in Ocular Microsurgery: A Safety and Workflow Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Tommy Korn, MD, Ophthalmologist - Sharp Rees-Stealy Medical Group, Sharp HealthCare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Spatial Ocular Microsurgery
Record Dates: First submitted 2025-12-06; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cataract Surgery; Cataract
Keywords: ocular microsurgery; spatial computing; eye surgery; Cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: The primary purpose of this study is to evaluate the safety and workflow impact of adjunctive head-mounted spatial computing visualization during standard-of-care ocular microsurgery. All enrolled participants undergo standard-of-care ocular microsurgery with adjunctive use of a head-mounted spatial computing visualization device. There is no comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Spatial computing visualization of cataract and anterior segment eye surgery (Experimental): Participants undergo standard-of-care cataract or anterior segment ocular surgery with adjunctive use of head-mounted spatial computing visualization. There is no comparison group.
  Interventions: Device: Apple Vision Pro (Head-Mounted Spatial Computing Display); Device: Zeiss Artevo Digital Surgical Microscope

INTERVENTIONS:
Device: Apple Vision Pro (Head-Mounted Spatial Computing Display) — Head-mounted spatial computing display used by the surgeon to view the real-time video output from the Zeiss Artevo digital surgical microscope. The Apple Vision Pro functions solely as an alternative visualization interface and does not acquire images, alter microscope function, modify surgical technique, or affect patient care.
Device: Zeiss Artevo Digital Surgical Microscope — FDA-cleared digital ophthalmic surgical microscope used as standard of care to visualize the operative eye during cataract and anterior segment surgery. The microscope provides the primary intraoperative imaging source for all cases, regardless of visualization display method.

SUMMARY:
The purpose of this research is to evaluate the use of the research study device, the Apple Vision Pro head-mounted spatial computing display, with the Zeiss Artevo 850 digital microscope system, for the visualization during cataract and anterior segment surgery. Specifically, researchers will assess how the study device affects surgical staff experience and workflow and monitor for patient safety and intraoperative complications associated with the use of the device.

DETAILED DESCRIPTION:
Surgeons and operating room staff will be asked to complete a survey regarding workflow, setup, and communication immediately after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled to undergo elective anterior segment eye surgery, including: cataract surgery, pterygium excision, corneal epithelial polishing
* Able and willing to provide informed consent prior to participation.

Exclusion Criteria:

* Complex ocular pathology that could interfere with surgical visualization or increase procedural risk, including but not limited to:
* Lens zonular instability or phacodonesis
* Prior vitreoretinal surgery (e.g., vitrectomy, scleral buckle, glaucoma drainage device) in the operative eye
* Significant corneal scarring, opacity, or edema
* Active ocular surface inflammation or infection
* Cognitive impairment or language barriers that prevent the patient from understanding and signing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative safety during head-mounted spatial computing visualization | Perioperative
  Safety will be assessed by the proportion of surgical cases completed using head-mounted spatial computing visualization without conversion to standard microscope visualization due to device-related issues, and by the occurrence of intraoperative complications potentially related to visualization, including posterior capsule rupture, vitreous loss, corneal or scleral injury, or other unplanned intraoperative events.

SECONDARY OUTCOMES:
Surgeon workload during ocular surgery | Immediately after surgery
  Surgeon workload measured using the National Aeronautics and Space Administration Task Load Index (NASA-TLX) questionnaire completed by the operating surgeon.
Surgeon-reported visualization quality and ergonomics | Immediately after surgery
  Surgeon-reported assessment of visualization clarity, comfort, ergonomic strain, and overall usability using a post-procedure survey.
Operating room staff workflow and usability | Immediately after surgery
  Operating room staff perception of workflow, communication, setup efficiency, and usability assessed using a post-procedure survey.
Operative time and setup efficiency | Perioperative
  Total operative time and setup duration recorded from the electronic medical record and intraoperative documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Korn, MD, Principal Investigator — Sharp Rees-Stealy Medical Group and Sharp HealthCare
Locations (1):
- Sharp HealthCare, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect patient confidentiality. Only aggregated, de-identified data will be published in scientific reports on visualization performance, workflow, and surgeon and operating room staff feedback.

REFERENCES:
- [Background] Brooke, J. (1996). SUS: A quick and dirty usability scale. In P. W. Jordan, B. Thomas, B. A. Weerdmeester, & I. L. McClelland (Eds.), Usability Evaluation in Industry (pp. 189-194). London: Taylor & Francis.
- [Background] Hart, S. G., & Staveland, L. E. (1988). Development of NASA-TLX (Task Load Index): Results of empirical and theoretical research. In P. A. Hancock & N. Meshkati (Eds.), Human Mental Workload (pp. 139-183). Amsterdam: North-Holland.
- [Background] Mastropasqua R, Ruggeri ML, Quarta A, Tartaro R, Vecchiarino L, Corboli LV, Brescia L, Orione M, Russo A, Avitabile T, Mastropasqua L. New Mixed Reality Headset: First Exploratory Use in Intraocular Surgery and Telementoring. Ophthalmol Ther. 2025 Jul;14(7):1597-1609. doi: 10.1007/s40123-025-01117-y. Epub 2025 Apr 11. PMID 40214829
- [Background] Broderick RC, Spurzem GJ, Jeffery Reeves J, Hollandsworth HM, Sandler BJ, Jacobsen GR, Longhurst CA, Horgan S. First use of augmented reality headset in minimally invasive general surgery: seeing is believing. Surg Endosc. 2025 Sep;39(9):6055-6060. doi: 10.1007/s00464-025-11985-x. Epub 2025 Jul 10. PMID 40640628
- [Background] Suh Y, Shin S, Kim BY, Jeong J, Kim TI. Comparison of neck angle and musculoskeletal discomfort of surgeon in cataract surgery between three-dimensional heads-up display system and conventional microscope. Sci Rep. 2024 Sep 30;14(1):22681. doi: 10.1038/s41598-024-68630-1. PMID 39349516